CLINICAL TRIAL: NCT02761252
Title: Bilastine and Montelukast in Patients With Seasonal Allergic Rhinoconjunctivitis and Asthma: Efficacy of Concomitant Administration - the SKY Study
Brief Title: Efficacy of Co-administration of Bilastine and Montelukast in Patients With SARC and Asthma
Acronym: SKY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Menarini International Operations Luxembourg SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEIN/15/Bil-ARC/001; 2015-004806-40 (EudraCT Number)
Record Dates: First submitted 2016-04-28; First posted 2016-05-04 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-04

CONDITIONS: Seasonal Allergic Rhinoconjunctivitis; Asthma
Keywords: Bilastine; Montelukast; total symptom score; AQLQ
MeSH Terms: conditions — Asthma | interventions — bilastine; montelukast

STUDY DESIGN:
Intervention Model Description: The study was a randomised (1:1:1), double-blind, double-dummy, interventional, active-controlled, parallel groups (three groups), multi-centre, multi-national, superiority clinical trial. The study plan included a 7-day (± 4) run-in period to ensure wash-out from previous forbidden treatments and to perform the tests required to ensure appropriate patient enrolment into the study. The active treatment period was 12 weeks (85 days) with a follow-up visit (phone call) at 28 days (± 4) after the End of Treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The principal investigator and study staff, subjects and monitors remained blinded to the treatment until study closure in this double-blind, double-dummy study. The identity of the study drug was revealed only if the subject experienced a medical emergency the management of which would be improved by the knowledge of the blinded treatment assignment.
  As the combination therapy of Bilastine + Montelukast consisted of two tablets in contrast to monotherapy with either Bilastine or Montelukast, the double-dummy technique was applied with matching placebo for each Investigation Medicinal Product (IMP) (monotherapy with Bilastine or Montelukast) to ensure the maintenance of double-blind conditions. Therefore, each patient took 2 tablets with each dose administered.
  As by randomisation list, each Patient Kit consisted of two IMP treatments (either active + placebo or active + active) in separate blisters packed in two different boxes.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bilastine+montelukast (Experimental): Bilastine 20 mg, 10 blister containing 10 tablets + Montelukast 10 mg, 10 blister containing 10 film coated tablets each for treatment
  Interventions: Drug: Bilastine 20mg; Drug: Montelukast 10mg
- Bilastine+placebo montelukast (Active Comparator): Bilastine 20 mg, 10 blister containing 10 tablets + Placebo Montelukast, 10 blister containing 10 film coated tablets each.
  Interventions: Drug: Bilastine 20mg; Drug: Placebo Montelukast 10mg
- Montelukast+placebo bilastine (Active Comparator): Placebo Bilastine, 10 blister containing 10 tablets + Montelukast 10 mg, 10 blister containing 10 film coated tablets each.
  Interventions: Drug: Montelukast 10mg; Drug: Placebo Bilastine 20mg

INTERVENTIONS:
Drug: Bilastine 20mg
  Other Names: Robilas
  Arms: Bilastine+montelukast; Bilastine+placebo montelukast
Drug: Montelukast 10mg
  Other Names: Montelukast
  Arms: Bilastine+montelukast; Montelukast+placebo bilastine
Drug: Placebo Bilastine 20mg
  Other Names: Placebo Bilastine
  Arms: Montelukast+placebo bilastine
Drug: Placebo Montelukast 10mg
  Other Names: Placebo Montelukast
  Arms: Bilastine+placebo montelukast

SUMMARY:
The purpose of this study is to compare concomitant administration of Montelukast and Bilastine to Montelukast and Bilastine monotherapies in patients with SARC and asthma

DETAILED DESCRIPTION:
The present study (SKY) was designed to show if once daily oral combination therapy with Montelukast 10 mg and Bilastine 20 mg is superior to monotherapy with Bilastine 20 mg in patients with Seasonal Allergic RhinoConjunctivitis (SARC) and comorbid mild to moderate asthma on total symptom scores (TSS) and if the combination therapy reflects an improvement in quality of life as assessed via the Asthma Quality of Life Questionnaire (AQLQ) over a longer time period when compared to monotherapies with Montelukast 10 mg and Bilastine 20 mg. Mild to moderate asthma was defined according to the criteria of the Global Initiative for Asthma, i.e., GINA criteria 2 and 3 (GINA, 2012). The study population included patients inadequately controlled on inhaled corticosteroids and in whom "as-needed" short acting beta-agonists provided inadequate clinical control.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients aged 18 years or older;
2. Patients with at least 2 years history of SARC prior to the study and mild to moderate asthma (GINA criteria 2 and 3) inadequately controlled on inhaled corticosteroids and in whom "as-needed" short acting beta-agonists provide inadequate clinical control;
3. Forced expiratory volume at one second (FEV1) > 70% of the predicted normal value demonstrable at least 6 hours after last short acting β-2 agonist use or 12 hours after last long acting β-2 agonist (LABA) use;
4. Nasal Symptoms Score (NSS) at baseline ≥ 3. Baseline NSS will be defined as the mean of the 6 last assessments of the patients' diary (3 last days before randomization);
5. Positive results of skin prick test on at least one seasonal allergen within the last 3 years;
6. Patients who provided a signed written informed consent form;
7. Patients who are able and willing to complete web-based Patient's Diary;
8. Patients who agree to maintain consistency in their surroundings throughout the study period;
9. Women of childbearing potential (WOCBP) including peri-menopausal women who have had a menstrual period within 1 year have to have a negative pregnancy test. Results have to be available until the Visit 2 and negative for the patient to be entered in the study.
10. WOCBP have to use an effective method of birth control throughout the study period and for 4 weeks after study completion (defined as a method which results in a failure rate of less than 1% per year) such as:

    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
    * progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
    * intrauterine device (IUD)
    * intrauterine hormone-releasing system (IUS)
    * bilateral tubal occlusion
    * vasectomised partner (provided that partner is the sole sexual partner of the trial participant and that the vasectomised partner has received medical assessment of the surgical success)
    * sexual abstinence In each case of delayed menstrual period (over one month between menstruations) confirmation of absence of pregnancy is strongly recommended. This recommendation also applies to WOCBP with infrequent or irregular menstrual cycles.

EXCLUSION CRITERIA

1. Patients with hypersensitivity to any component of the study medications;
2. Patients with non-allergic rhinoconjunctivitis (e.g. vasomotor, infectious, drug-induced);
3. Presence of nasal polyps or any clinically important nasal anomaly;
4. History of acute and/or chronic sinusitis within 30 days of Visit 2;
5. History of eye surgery within 3 months of Visit 2;
6. History of intranasal surgery within 3 months of Visit 2;
7. Immunotherapy within 6 months prior to Visit 1;
8. Upper respiratory infections including cold and systemic infections within 3 weeks of Visit 2;
9. Patients with moderate to severe renal impairment and taking P-gp inhibitors (e.g. ketoconazole, erythromycin, cyclosporine, ritonavir, diltiazem) within 7 days prior to the first dose of study medication;
10. Patients requiring daily "controller" medications with cromolyn-type drugs or leukotriene antagonists;
11. Patient required daily "controller" medication with Inhaled corticosteroids (ICS) or LABA at medium /high dosage defined by GINA criteria;
12. Patients with clinically important (based on principal investigator's judgment) hepatic impairment;
13. Patients with severe concomitant disease (based on principal investigator's judgment) that could interfere with treatment response;
14. Patients with QT syndrome;
15. Patients with Galactose intolerance, Lapp lactase deficiency or glucose- galactose malabsorption;
16. Pregnant or breast-feeding women;
17. Patients with a mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study (based on principal investigator's judgment);
18. Patients who had a recent history (within previous 12 months) of drug addiction or alcohol abuse based on Principal investigator's judgment ;
19. Patients participating in or having participated in another clinical trial within the previous three months;
20. Patients unable to take relief medications due to contraindications or intolerance;
21. Patients who are taking or have taken any of the following medications prior to randomisation in the study and have not complied with the specified washout period:

    * Antihistaminic drugs or montelukast (7 days)
    * Systemic or intranasal corticosteroids (4 weeks)
    * Delayed-release corticosteroids (3 months)
    * Ketotifen (2 weeks)
    * Macrolides antibiotics and imidazolic antifungals (systemic)(7 days)
    * Anticholinergics (7 days)
    * Drugs with antihistamine properties (phenothiazine) (7 days)
    * Intranasal and systemic decongestants (3 days)
    * Lodoxamide (7 days)
22. Patients who will be operating heavy machinery or need to drive motor vehicles as an essential part of their profession.
23. Patients who are planning to travel outside the study area during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Pistolesi, Prof, Study Director — AOUC Azienda Ospedaliero-Universitaria Careggi; Oliviero Rossi, Prof, Study Director — AOUC Azienda Ospedaliero-Universitaria Careggi
Locations (32):
- Croatia (3):
  - Čakovec
  - Rijeka
  - Zagreb
- Czechia (3):
  - Brno
  - Ostrava Hrabuvka
  - Teplice
- Germany (2):
  - Dreieich
  - Heidelberg
- Italy (5):
  - Catania
  - Florence
  - Modena
  - Pavia
  - Verona
- Riga, Latvia
- Poland (12):
  - Bialystok
  - Bielsko-Biala
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Nowy Duninów
  - Poznan
  - Rzeszów
  - Tarnów
  - Wroclaw
- Romania (4):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Ploieşti
- Slovakia (2):
  - Bardejov
  - Levice

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started on 13 April 2016 and termineted on 23 November 2016. 454 patients with SARC and mild to moderate asthma as comorbidity were screened.
  420 patients were randomised of which 388 patients completed the study.
Pre-assignment Details: 454 patients were enrolled but 34 patients did not met inclusion/exclusion critera.
Groups:
- Bilastine+Montelukast: Bilastine 20mg
  Montelukast 10mg
- Bilastine Monotherapy: Bilastine 20mg
  Placebo Montelukast 10mg
- Montelukast Monotherapy: Montelukast 10mg
  Placebo Bilastine 20mg
Period: Overall Study
Arm/Group | Bilastine+Montelukast | Bilastine Monotherapy | Montelukast Monotherapy
Started | 143 | 140 | 137
Completed | 133 | 132 | 123
Not Completed | 10 | 8 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bilastine+Montelukast | Bilastine Monotherapy | Montelukast Monotherapy | Total
Number analyzed (Participants) | 143 | 140 | 137 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 143 | 140 | 137 | 420
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (11.1) | 35.5 (11.0) | 35.4 (10.7) | 35.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 83 | 73 | 225
  Male | 74 | 57 | 64 | 195

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline With Montelukast+Bilastine Compared With Bilastine Monotherapy in SARC Symptoms
Description: To demonstrate that concomitant administration of montelukast and bilastine is superior to bilastine monotherapy in SARC symptoms, as assessed by Total Symptoms Scores (TSS) after 4 weeks of treatment.
  Total Symptoms Scores (TSS) assesses nasal (nasal congestion, rhinorrhea, nasal itching, sneezing) and non nasal symptoms (ocular redness, ocular itching, tearing) of rhinoconjuctivits.
  Each of the 7 symptoms is scored from 0 (absent) to 3 (severe) as follows:
  * 0 (absent) Symptom not present
  * 1 (mild) Symptom is clearly present but easily tolerated, a nuisance, minimal awareness
  * 2 (moderate) Symptom is bothersome but tolerable, does not interfere with daily activities or sleep
  * 3 (severe) Symptom is hard to tolerate and interferes with daily activities or sleep.
  TSS assessment comprises of scoring (0-3) of all 7 above mentioned symptoms. Final TSS scores is in a range from 0-21.
Time Frame: 4 weeks of treatment (from baseline to 4 weeks of treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Bilastine+Montelukast: Bilastine 20mg+Montelukast 10mg
Arm/Group | Bilastine+Montelukast | Bilastine Monotherapy
Number analyzed (Participants) | 143 | 140
score on a scale | -3.2522 [-3.8718 to -2.6327] | -3.4462 [-4.0708 to -2.8217]
Statistical Analysis 1: Comparison: Bilastine+Montelukast vs Bilastine Monotherapy; Test type: Superiority; p = 0.5721, ANCOVA; Mean Difference (Final Values) = -0.194, 95% CI 2-sided [-0.8693 to 0.4813], Standard Error of Mean 0.3429

2. Secondary Outcome: Change From Baseline With Montelukast+Bilastine Compared With Montelukast and Bilastine Monotherapies in Asthma Control
Description: To evaluate the efficacy of concomitant montelukast and bilastine compared with montelukast and bilastine monotherapies in asthma control, as assessed by Asthma Quality of Life Questionnaire (AQLQ) after 4 weeks.
  The AQLQ was developed to measure the functional problems (physical, emotional, social and occupational) that are most troublesome to adults (17-70 years) with asthma.
  Each of the 32 questionnaire's items will be scored on a 7-point scale (where 7 means "not impaired at all" and 1 means "severely impaired"). The overall AQLQ score is the mean of all 32 responses (https://www.qoltech.co.uk/aqlq.html).
  The change in AQLQ score from baseline to 4 weeks after treatment - AQLQ score at baseline for patients with both available values has been the secondary endpoint.
Time Frame: After 4 weeks of treatments
Population: The Intention To Treat population (used for statistical analysis) was 419 patients because 1 patient in Montekukast Monotherapy arm was a drop-out.
  The drop-out patient was, instead, included in a Safety Population (420 patients).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Bilastine+Montelukast: Bilastine 20mg + Montelukast 10mg
Arm/Group | Bilastine+Montelukast | Bilastine Monotherapy | Montelukast Monotherapy
Number analyzed (Participants) | 143 | 140 | 136
score on a scale | 0.6250 [0.4788 to 0.7712] | 0.6399 [0.4929 to 0.7870] | 0.5849 [0.4344 to 0.7353]
Statistical Analysis 1: Comparison: Bilastine+Montelukast vs Bilastine Monotherapy vs Montelukast Monotherapy; Test type: Superiority; p = 0.0105, ANCOVA; Mean Difference (Final Values) = -1.1552, 95% CI 2-sided [-2.0379 to -0.2725], Standard Error of Mean 0.4489

3. Secondary Outcome: Change From Baseline With Montelukast+Bilastine Compared With Montelukast and Bilastine Monotherapies in SARC Symptoms (DNSS)
Description: To evaluate the efficacy of concomitant montelukast and bilastine compared with montelukast and bilastine monotherapies in daytime symptoms of SARC, as assessed by Daytime Nasal Symptom Score (DNSS) after 4 weeks of treatment.
  Daytime Nasal Symptom Score (DNSS) is the average of individual scores of nasal congestion, rhinorrhea, nasal itching, sneezing of rhinoconjuctivits.
  Each of the 4 symptoms is scored from 0 (absent) to 3 (severe) as follows:
  * 0 (absent) Symptom not present
  * 1 (mild) Symptom is clearly present but easily tolerated, a nuisance, minimal awareness
  * 2 (moderate) Symptom is bothersome but tolerable, does not interfere with daily activities or sleep
  * 3 (severe) Symptom is hard to tolerate and interferes with daily activities or sleep.
  DNSS assessment comprises of scoring (0-3) of all 4 above mentioned symptoms. Final DNSS scores is in a range from 0-12.
Time Frame: After 4 weeks of treatment (from baseline)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Bilastine+Montelukast | Bilastine Monotherapy | Montelukast Monotherapy
Number analyzed (Participants) | 143 | 140 | 136
score on a scale | -1.9713 [-2.3442 to -1.5984] | -2.1106 [-2.4863 to -1.7349] | -1.8678 [-2.2468 to -1.4888]
Statistical Analysis 1: Comparison: Bilastine+Montelukast vs Bilastine Monotherapy vs Montelukast Monotherapy; Test type: Superiority; p = 0.4885, ANCOVA; Mean Difference (Final Values) = -0.1393, 95% CI 2-sided [-0.5342 to 0.2557], Standard Error of Mean 0.2009

4. Secondary Outcome: Change From Baseline With Montelukast + Bilastine Compared With Montelukast and Bilastine Monotherapies in SARC Symptoms (DNNSS)
Description: To evaluate the efficacy of concomitant montelukast and bilastine compared with montelukast and bilastine monotherapies in daytime symptoms of SARC, as assessed by Daytime Non Nasal Symptom Score (DNNSS) after 4 weeks of treatment.
  Daytime Non Nasal Symptom Score (DNSS) is the average of individual scores of ocular redness, ocular itching and tearing of rhinoconjuctivits.
  Each of the 3 symptoms is scored from 0 (absent) to 3 (severe) as follows:
  * 0 (absent) Symptom not present
  * 1 (mild) Symptom is clearly present but easily tolerated, a nuisance, minimal awareness
  * 2 (moderate) Symptom is bothersome but tolerable, does not interfere with daily activities or sleep
  * 3 (severe) Symptom is hard to tolerate and interferes with daily activities or sleep.
  DNNSS assessment comprises of scoring (0-3) of all 3 above mentioned symptoms. Final DNNSS scores is in a range from 0-9.
Time Frame: After 4 weeks of treatment (from baseline)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Bilastine+Montelukast | Bilastine Monotherapy | Montelukast Monotherapy
Number analyzed (Participants) | 143 | 140 | 136
score on a scale | -1.2824 [-1.5667 to -0.9980] | -1.3185 [-1.6051 to -1.0320] | -1.1574 [-1.4462 to -0.8687]
Statistical Analysis 1: Comparison: Bilastine+Montelukast vs Bilastine Monotherapy vs Montelukast Monotherapy; Test type: Superiority; p = 0.81032, ANCOVA; Mean Difference (Final Values) = -0.03615, 95% CI 2-sided [-0.3319 to 0.2596], Standard Error of Mean 0.1504

5. Secondary Outcome: Usage of Relief Medication for SARC
Description: Number of days without any relief medication for SARC
Time Frame: From baseline to 4 weeks of treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Bilastine+Montelukast | Bilastine Monotherapy | Montelukast Monotherapy
Number analyzed (Participants) | 143 | 140 | 136
Days | 15.0057 (0.8260) | 15.8416 (0.8326) | 15.4179 (0.8411)
Statistical Analysis 1: Comparison: Bilastine+Montelukast vs Bilastine Monotherapy vs Montelukast Monotherapy; Test type: Other; p = 0.3704, ANOVA; Mean Difference (Final Values) = 0.8359, 95% CI 2-sided [-0.9969 to 2.6688], Standard Error of Mean 0.9322

6. Secondary Outcome: Usage of Relief Medication for Asthma
Description: Number of days without any relief medication for Asthma.
Time Frame: From baseline to 4 weeks of treatment
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Bilastine+Montelukast | Bilastine Monotherapy | Montelukast Monotherapy
Number analyzed (Participants) | 143 | 140 | 136
Days | 53.2548 (2.0193) | 52.4177 (2.0212) | 50.7146 (2.0768)
Statistical Analysis 1: Comparison: Bilastine+Montelukast vs Bilastine Monotherapy vs Montelukast Monotherapy; Test type: Superiority; p = 0.7452, ANOVA; Median Difference (Final Values) = -0.837, 95% CI 2-sided [-5.8968 to 4.2228], Standard Error of Mean 2.5735

ADVERSE EVENTS:
Groups:
- Bilastine+Montelukast: Bilastine 20 mg, 10 blister containing 10 tablets + Montelukast 10 mg, 10 blister containing 10 film coated tablets each for treatment
  Bilastine 20mg
  Montelukast 10mg
- Bilastine+Placebo Montelukast: Bilastine 20 mg, 10 blister containing 10 tablets + Placebo Montelukast, 10 blister containing 10 film coated tablets each.
  Bilastine 20mg
  Placebo Montelukast 10mg
- Montelukast+Placebo Bilastine: Placebo Bilastine, 10 blister containing 10 tablets + Montelukast 10 mg, 10 blister containing 10 film coated tablets each.
  Montelukast 10mg
  Placebo Bilastine 20mg
Arm/Group | Bilastine+Montelukast | Bilastine+Placebo Montelukast | Montelukast+Placebo Bilastine
Serious Adverse Events (participants affected / at risk) | 0/143 | 0/140 | 1/137
Other Adverse Events (participants affected / at risk) | 8/143 | 4/140 | 14/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilastine+Montelukast (N=143) | Bilastine+Placebo Montelukast (N=140) | Montelukast+Placebo Bilastine (N=137)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilastine+Montelukast (N=143) | Bilastine+Placebo Montelukast (N=140) | Montelukast+Placebo Bilastine (N=137)
Alanine Aminotransferase Increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamytrasferase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes